CLINICAL TRIAL: NCT00403858
Title: A Single Centre Study to Assess the Safety and Efficacy of Movicol in the Treatment of Faecal Impaction in Children Followed by a Double Blind, Randomised Phase to Compare the Safety and Efficacy of Movicol and Lactulose for Maintenance Therapy
Brief Title: Movicol in Childhood Constipation (ProMotion Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99/05 (Part I)
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2007-01

CONDITIONS: Feces, Impacted
MeSH Terms: conditions — Fecal Impaction | interventions — Lactulose

INTERVENTIONS:
Drug: Polyethylene glycol 3350 NA bicarbonate NaCl KCl (Movicol)
Drug: Lactulose

SUMMARY:
This was a single centre study comprised of two stages (Parts I and II). Part I was a 9-day open label evaluation of Movicol administered to patients in hospital. This study evaluated the safety and efficacy of Movicol in treating faecal impaction. Movicol was administered over 3 - 7 days to achieve disimpaction.

DETAILED DESCRIPTION:
Patients received Movicol treatment until disimpaction was achieved according to the following regime:

Day 1: Ages 2 - 4 received 1 (one) sachet whilst 5 - 11 year olds received 2 (two).

Day 2: Ages 2 - 4 received 2 (two) sachets whilst 5 - 11 year olds received 3 (three).

Day 3: Ages 2 - 4 received 2 (two) sachets whilst 5 - 11 year olds received 4 (four).

Day 4: Ages 2 - 4 received 3 *three) sachets whilst 5 - 11 year olds received 5 (five).

Day 5: Ages 2 - 4 received 3 (three) sachets whilst 5 - 11 year olds received 6 (six).

Day 6: Ages 2 - 4 received 4 (four) sachets whilst 5 - 11 year olds received 6 (six).

Day 7: Ages 2 - 4 received 4 (four) sachets whilst 5 - 11 year olds received 6 (six).

If on day 8 the patient was still impacted they were withdrawn from study and treated according to their individual needs. Disimpaction was assessed clinically (loss of faecal masses and passage of watery stools).

Two days following disimpaction patients were randomised (according to the randomisation list) to receive Movicol or Lactulose Dry. During bowel retraining the appropriate maintenance dose of Movicol or Lactulose Dry was determined. Patients were discharged once they were passing regular, painless, bowel actions.

ELIGIBILITY:
Inclusion Criteria:

* patients that, in the opinion of the investigator, are constipated/fecally impacted as to require hospital stay to treat and/or relieve the impaction
* children aged 2 - 11 years old inclusive
* patients of either sex

Exclusion Criteria:

Patients with

* intestinal perforation or obstruction
* severe inflammatory conditions of the intestinal tract
* uncontrolled renal/hepatic/cardiac diseases
* uncontrolled endocrine disorder(s)
* any neuromuscular condition affecting bowel function
* hypersensitivity to lactulose or PEG or other constituent of Movicol
* patients who have taken any investigational drug in the three months
* patients or patients whose parents would in the opinion of the investigator are unable to comply with requirements of the study

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2000-10; Study Completion 2002-04

PRIMARY OUTCOMES:
evaluate the safety and efficacy of Movicol in the treatment of faecal impaction in children.

CONTACTS AND LOCATIONS:
Overall Officials: David CA Candy, MD, Principal Investigator — St. Richard's Hospital
Locations (1):
- St Richard's Hospital, Royal West Sussex Hospital NHS Trust, Chichester, United Kingdom

REFERENCES:
- [Background] Dalziel SR et al. Efficacy of Movicol in children with faecal impaction. A series of en case histories (A13). British Society of Paediatric Gastroenterologists Annual Meeting. Bristol:21-22, Jan 2000
- [Background] Attar A, Lemann M, Ferguson A, Halphen M, Boutron MC, Flourie B, Alix E, Salmeron M, Guillemot F, Chaussade S, Menard AM, Moreau J, Naudin G, Barthet M. Comparison of a low dose polyethylene glycol electrolyte solution with lactulose for treatment of chronic constipation. Gut. 1999 Feb;44(2):226-30. doi: 10.1136/gut.44.2.226. PMID 9895382
- [Result] Candy DC, Edwards D, Geraint M. Treatment of faecal impaction with polyethelene glycol plus electrolytes (PGE + E) followed by a double-blind comparison of PEG + E versus lactulose as maintenance therapy. J Pediatr Gastroenterol Nutr. 2006 Jul;43(1):65-70. doi: 10.1097/01.mpg.0000228097.58960.e6. PMID 16819379